CLINICAL TRIAL: NCT07347912
Title: Group-based Resistance Training for Adults With Down Syndrome; a Feasibility Pilot Randomised Control Crossover Trial
Brief Title: Group-based Resistance Training for Adults With Down Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John of God Intellectual Disability Services - Dublin South East (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Sharon Hardiman, Senior Clinical Psychologist, Saint John of God Intellectual Disability Services - Dublin South East
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ID2046
Record Dates: First submitted 2025-11-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome; Healthy Aging; Resistance Training
Keywords: Dementia Risk Reduction; Proactive Intervention
MeSH Terms: conditions — Down Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a pilot randomised control crossover trial study that will use a mixed methods approach to assess the feasibility and efficacy of group based resistance training (RT) for adults with Down syndrome attending a community based intellectual disability service. To mitigate the potential limitations of a small sample size, a crossover design will be employed meaning participants initially assigned to the services as usual control group will become experimental participants (and take part in the RT programme), after the first intervention group have completed their 3-month follow-up assessment. Accordingly, after the crossover, participants originally allocated to the experimental group will attend the remaining assessment sessions as services as usual participants.
Who Masked: Outcomes Assessor
Masking Description: Efficacy data will be collected by the Research Assistant who will be blind to group membership. The Efficacy data will be anonymized by removal of any directly identifying component and the pseudonymizing "key" will be held by the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training (Experimental): Individuals in this group will initially attend the 12-week (24 session) RT programme. They will also attend assessment sessions at baseline, post-programme and three-month follow-up. After the crossover, the experimental group will receive their services as usual and attend the remaining assessment sessions (post-programme; three-month follow-up) as control participants.
  Interventions: Behavioral: Resistance Training
- Services as Usual Control Group (Other): Individuals in the services as usual control group will initially attend their services as usual for 12 weeks. They will also attend assessment sessions at baseline, post-programme and three-month follow-up. After the crossover, the services as usual control group will receive the 12-week (24 session) RT programme and will attend remaining assessment sessions (post-programme; three-month follow-up) as experimental participants.
  Interventions: Other: Services as Usual Control Group

INTERVENTIONS:
Behavioral: Resistance Training — Resistance Training (or RT for short) is a popular form of physical exercise, which focuses on improving muscle strength and endurance using weighted or resistance-based exercises.
  RT can involve 'lifting weights', doing resistance band movements or performing bodyweight exercises.
  Arms: Resistance Training
Other: Services as Usual Control Group — Participants will receive services as usual for the initial 12-week period prior to crossover to the resistance training intervention. During Period 2 (12 weeks), participants initially assigned to the resistance training group return to services as usual control group.
  Arms: Services as Usual Control Group

SUMMARY:
The investigators are interested in Resistance Training as a physical exercise intervention for adults with Down syndrome. Resistance Training (or RT for short) is a popular form of physical exercise, which focuses on improving muscle strength and endurance using weighted or resistance-based exercises. RT can involve 'lifting weights', doing resistance band movements or performing bodyweight exercises. Researchers have developed a tailored programme of RT exercises (called RESID), which are suitable and safe to implement for individuals with mild to moderate intellectual disabilities. RT has been shown to help people improve thinking skills and overall quality of life. RT has been associated with better brain health in older adults with memory problems. The investigators want to run the RESID exercise programme with adults with Down syndrome who do not have memory problems but who the investigators know are at much greater risk of developing memory problems as they get older. The investigators are hoping this programme will support brain health and healthy ageing in adults with Down syndrome. The investigators want to see this programme can be successfully run with people with intellectual disabilities. The investigators want to see if participants enjoy this programme and engage well with it. The investigators want to see if there are any barriers to participating in this programme. The investigators also want to see how much it will cost to run this programme again in the future. The investigators also want to see if this programme helps these adults to feel better about themselves, to have better memory skills, to have better day-to-day skills, and to have better strength and mobility. The investigators will measure study outcomes using self-report scales, a memory assessment, strength test, mobility tests, blood pressure/heart rate test and by getting information from caregivers. The investigators will use the same measures with a similar group of adults who initially do not take part in this programme. They will be called our services as usual control group. During the first group, these adults will attend usual weekly services. However, they will be offered a place on a RT programme after the first experimental group have finished. The investigators will decide the order of who takes part in which initial group (Experimental or Control) by drawing names out of a hat so that it will be as fair as possible. However, all participants in this study will eventually take part in the RT programme. The investigators hope this study will tell us a lot about running a RT programme for people with intellectual disabilities. The investigators hope the results of this research study will show that adults with Down syndrome enjoy and engage well with this programme and that RT has benefits for adults with Down syndrome who do not memory problems. The investigators hope to show that RT can support the healthy ageing of adults with Down syndrome.

DETAILED DESCRIPTION:
The proposed study intends to measure the feasibility and efficacy of a standardised group-based resistance training (RT) exercise program for adults with an intellectual disability (ID) at high risk of developing Alzheimer's disease (AD) in the future. Adults with Down syndrome (DS) are at "ultra-high" risk of developing AD as they age. However, there is a dearth of research studies focusing on brain health strategies for this population. Physical activity (PA) is emerging as key brain health booster. PA has been shown to affect brain plasticity influencing both cognition and well-being. Encouragingly, there is emerging evidence that PA can boost cognitive reserve in adults with DS. RT is a popular form of physical exercise, which focuses on improving muscle strength using weighted or resistance-based exercises. RT has been shown to be an important dementia risk-reduction strategy for adults in the general population. A standardised resistance exercise set for a total body workout for adults with mild or moderate intellectual disabilities (RESID) has recently been developed. The current research will focus on evaluating the benefits of this RESID programme for adults with DS who are at "ultra-high" risk of developing AD in the future. The study will be conducted as a pilot randomised control crossover trial with all participants eventually receiving the RT intervention. Study results will contribute significantly to our understanding of the impact of proactive RT on key health and well-being outcomes for adults with Down Syndrome.

The information collected in this study will be limited to the information that is needed to answer the research study questions. With the consent of participants, the investigators will seek to place some of the assessment information on participants' Clinical (Psychology) File. This information will be important for the person if there are concerns about memory/cognitive skills in the future. This information will be stored safely on the Psychology File and will only be accessed by the Psychology Team. The investigators will also seek to deposit the anonymous data from this study in a secure anonymous data register for future research projects but only where these projects are approved by a Research Ethics Committee. With the participants' consent, the investigators will seek to deposit an anonymous data file derived from this study in a secure anonymous future Saint John of God Data register by the year 2034 to be used for future research projects but only where these projects are approved by a Research Ethics Committee. This data register has not yet been built but the investigators want to fully inform the potential participants of what will happen to the anonymous data derived from personal data.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Previous diagnosis of Down Syndrome;
* Previous diagnosis of Mild to Moderate Intellectual Disability;
* Aged between 20 to 45 years old;
* Capable of providing consent to participate in this research study;
* Have a close caregiver (proxy participant) who also consents to take part in this study.

Proxy:

* Be a close caregiver (family or staff) for a participant;
* Consent to participate in this research study.

Exclusion Criteria:

Participants:

* Severe or Profound Intellectual Disability;
* Significant behaviours of concern that would preclude group participation;
* Showing signs of dementia at pre-screening (on the G-DSDS);
* does not have a close caregiver who consents to take part in this study.

Proxy:

* none

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Episodic Memory | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Episodic Memory will be assessed using The FULD Object Memory Evaluation Test (FOME) which is a published standardized test. This test will be individually administered to each participant by the Research Assistant (RA) during their assessment sessions. The FOME has been found to be a reliable and valid measure of episodic memory (with reliability coefficients ranging from 0.91 to 0.96). It evaluates the episodic memory functions of encoding, storage, and recall across five recall trials (score range 0 to 50; higher scores indicating greater episodic memory) and a delayed recall trial (score range 0 to 10; higher scores indicating greater episodic memory). This scale will be completed by the participant during their assessment sessions with the RA. It is estimated that this measure will take about 10 minutes to complete.
Adaptive Behaviour | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Adaptive Behaviour will be measured using the Vineland Adaptive Behaviour Scales (3rd Edition). The Domain-Level Parent/Caregiver Form will be completed by Proxy participants during each assessment period. The Vineland Adaptive Behaviour Scales is a valid and reliable (Cronbach alpha scores range from 0.93 to 0.97) measure of personal and social skills needed for everyday living. It is widely used to assess the adaptive behaviour of adults with intellectual disabilities. It provides three standardised domain scores: communication (standard score range 20 to 140; higher scores indicating better communication), socialisation (standard score range 20 to 140; higher scores indicating better socialisation), and daily living skills (standard score range 20 to 140; higher scores indicating better daily living skills) and an overall adaptive behaviour composite score (standard score range 20 to 140; higher scores indicating better adaptive behavior. It takes about 10 - 15 minutes to complete.
Grip Strength | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Grip strength will be measured using a handheld Jamar® Smart Hand Dynamometer, an established tool for evaluating isometric grip force. Assessment will be administered by a registered Physiotherapist at SJOG-DSE. Estimated duration: <5 minutes. Unit of Measure: Kilograms of force (kg). The higher the kg or force, the stronger the grip.
Mobility | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Mobility will be assessed using the Timed Up and Go (TUG) test, which measures the time taken to stand up from a chair, walk 3 meters, turn, walk back, and sit down. Administered by a registered Physiotherapist. Estimated duration: <5 minutes. Unit of Measure: Seconds (s).
Leg Strength | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Mobility will also be assessed using the Sit to Stand test, which measures the number of times a participant can rise from a chair to a full standing position within 30 seconds. Assessment will be administered by a registered Physiotherapist. Estimated duration: <5 minutes. Unit of Measure: Number of repetitions in 30 seconds.
Blood Pressure | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Blood pressure will be measured using a calibrated sphygmomanometer in a seated position after 5 minutes rest. Blood pressure will be taken by a registered nurse. Estimated duration: <5 minutes. Unit of Measure: Millimeters of mercury (mmHg). A healthy blood pressure is below 120/80 mmHg.
Body Mass Index | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  BMI is a measurement of a person's leanness based on their height and weight, and is intended to quantify tissue mass. It is widely used as a general indicator of whether a person has a healthy body weight for their height. Specifically, the value obtained from the calculation of BMI is used to categorize whether a person is underweight, normal weight, overweight, or obese depending on what range the value falls between. Heigh (cm) and Weight (kg) will be measured by a healthcare professional. Unit of Measure: kg/m²
  Ranges:
  Underweight: BMI less than 18.5 kg/m². Normal weight: BMI between 18.5 and 24.9 kg/m². Overweight: BMI between 25 and 29.9 kg/m². Obese: BMI of 30 kg/m² or higher.
Resting Heart Rate | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Resting heart rate will be measured using a heart rate monitor after 5 minutes rest. This measure will be taken by a registered nurse. Estimated duration: <5 minutes. Unit of Measure: Beats per minute (bpm). A lower resting heart rate generally indicates better cardiovascular fitness and a more efficient heart. Regular exercise and physical activity can lead to a lower resting heart rate over time.
Attendance Rate | Across all sessions during the initial programme (24 sessions over 12 weeks) Across all sessions during the crossover programme (24 sessions over 12 weeks)
  Attendance will be recorded for each scheduled session. Unit of Measure: Percentage of sessions attended per participant
Session Satisfaction (Participant-Reported) | Immediately after each session throughout the programme (24 sessions over 12 weeks Immediately after each session in the crossover phase (24 sessions over 12 weeks)
  Participants will rate their satisfaction at the end of each session using an adapted "easy read" 5-point Likert scale (0 = "No!" to 5 = "Yes, a lot!"). Higher scores indicate greater satisfaction.
  Unit of Measure: Score on 0-5 Likert scale (higher = greater satisfaction)
Trainer-Reported Engagement Score | Time Frame: Immediately after each session throughout the programme (24 sessions over 12 weeks) Immediately after each session in the crossover phase (24 sessions over 12 weeks)
  Trainers will rate participant engagement across four domains: interest, communication, enjoyment, and mood. Each domain scored on a 0-4 scale. Higher ratings indicate more favorable interest, communication, enjoyment, and mood. Unit of Measure: Score per domain (0-4).
Resource Cost (Hours) | Through study completion (approximately 18 months)
  Total hours required for program adaptation, planning, delivery, and evaluation will be recorded. Unit of Measure: Hours.
Equipment costs in Euro € | Through study completion, approximately 18 months.
  Total cost of equipment required to run the RT program. Each item will be itemized and costed individually and then totaled. Unit of Measure: Cost in Euros €.
Recruitment Rate | Approximately 4-6 months recruitment period.
  Recruitment rate will be calculated as the proportion of participants recruited from the total eligible pool, along with the average monthly recruitment rate.
  Unit of Measure: Percentage of eligible participants recruited.
Retention Rate | Through study completion (approximately 18 months)
  Retention rate will be calculated as the number of individuals that completed the follow-up measures as a proportion of those recruited.
  Unit of Measure: Percentage of recruited participants completing all assessments.

SECONDARY OUTCOMES:
Subjective Wellbeing | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Subjective well-being will be measured using a measure called the Personal Well-Being Score (PWS). The PWS is a brief self-report measure of generic well-being developed for routine use in person-centred care and healthcare quality improvement. The PWS will be completed by the participant during their assessment session (pre-post-follow up) with the Research Assistant (RA). The PWS has been shown to have good psychometric properties (Cronbach's alpha > 0.80). Each of the four PWS items will be scored on a 5-point scale from 0 (Disagree a lot) to 4 (Agree a lot) with higher scores indicating greater subjective wellbeing. A PWS summary score will be calculated by adding scores across all four items (range 0 to 16; higher scores indicating better subjective wellbeing).
  It is estimated that this measure will take about 5 minutes to complete.
Memory Self-efficacy | Baseline (1-2 weeks pre program) Post (1-2 weeks post program) 3-month follow-up (12-14 weeks post-program) Crossover Baseline (1-2 weeks pre program) Crossover Post (1-2 weeks post program) Crossover 3-month follow-up (12-14 weeks post-program)
  Memory self-efficacy will be assessed using a self-rating scale developed by the Research Team. This scale will ask participants to rate their own memory in areas found to be most affected during early-stage dementia. Responses will be rated on a 5-point Likert scale (pictorially represented by faces and symbols to aid accessibility; range 0 "never" have difficulty to 4 "always" have difficulty in the past two months). Responses will be summed to provide a total score of 0 to 24 (0 = no memory difficulty reported to 24 = memory difficulties "always" in all areas measured). This scale will be completed by the participant during their assessment sessions with the RA. It is estimated that this measure will take about 15 minutes to complete.
Rate of Perceived Exertion - staff rated | Immediately after each exercise during each session throughout the programme (24 sessions over 12 weeks) Immediately after each exercise during each session in the crossover phase (24 sessions over 12 weeks)
  The modified Borg CR10 RPE scale measures exertion on a scale of 0 (no exertion or resting) to 10 (pushing yourself to the max). Staff will observe participant's level of exertion including breathing rate and breathlessness to determine the participant's RPE during each exercise during each session.
Adapted Rate of Perceived Exertion - participant self-rated | Immediately after each session throughout the programme (24 sessions over 12 weeks Immediately after each session in the crossover phase (24 sessions over 12 weeks)
  Participants will rate their level of perceived exertion at the end of each session using an adapted "easy read" 4-point Likert scale (0 = "little effort" to 4 = "the most effort"). Higher scores indicate higher effort.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hardiman, Principal Investigator — Saint John of God Intellectual Disability Services - Dublin South East
Locations (1):
- Saint John of God Intellectual Disability Services - Dublin South East, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costall B, Kelly ME, Naylor RJ. The antidyskinetic action of dihomo-gamma-linolenic acid in the rodent. Br J Pharmacol. 1984 Nov;83(3):733-40. doi: 10.1111/j.1476-5381.1984.tb16227.x. PMID 6542444
- [Background] Panel on Measuring Subjective Well-Being in a Policy-Relevant Framework; Committee on National Statistics; Division on Behavioral and Social Sciences and Education; National Research Council; Stone AA, Mackie C, editors. Subjective Well-Being: Measuring Happiness, Suffering, and Other Dimensions of Experience [Internet]. Washington (DC): National Academies Press (US); 2013 Dec 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK174473/ PMID 24432436
- [Background] Chung JC. Clinical validity of Fuld Object Memory Evaluation to screen for dementia in a Chinese society. Int J Geriatr Psychiatry. 2009 Feb;24(2):156-62. doi: 10.1002/gps.2085. PMID 18612999
- [Background] FULD, P.A. The Fuld Object Memory Evaluation. Chicago: Stoelting Instrument Company, 1981
- [Background] Sparrow, S. S., Cicchetti, D. V., & Saulnier, C. A. (2016). Vineland Adaptive Behavior Scales, Third Edition. Bloomington, MN: Pearson Assessment.
- [Background] Benson T, Sladen J, Liles A, Potts HWW. Personal Wellbeing Score (PWS)-a short version of ONS4: development and validation in social prescribing. BMJ Open Qual. 2019 Apr 11;8(2):e000394. doi: 10.1136/bmjoq-2018-000394. eCollection 2019. PMID 31206049
- [Background] Weinberg, R. S., & Gould, D. (2015). Foundations of sport and exercise psychology (6th ed.). Champaign, IL: Human Kinetics
- [Background] Pape SE, Baksh RA, Startin C, Hamburg S, Hithersay R, Strydom A. The Association between Physical Activity and CAMDEX-DS Changes Prior to the Onset of Alzheimer's Disease in Down Syndrome. J Clin Med. 2021 Apr 27;10(9):1882. doi: 10.3390/jcm10091882. PMID 33925348
- [Background] Ptomey LT, Szabo AN, Willis EA, Gorczyca AM, Greene JL, Danon JC, Donnelly JE. Changes in cognitive function after a 12-week exercise intervention in adults with Down syndrome. Disabil Health J. 2018 Jul;11(3):486-490. doi: 10.1016/j.dhjo.2018.02.003. Epub 2018 Feb 26. PMID 29501470
- [Background] Broadhouse KM, Singh MF, Suo C, Gates N, Wen W, Brodaty H, Jain N, Wilson GC, Meiklejohn J, Singh N, Baune BT, Baker M, Foroughi N, Wang Y, Kochan N, Ashton K, Brown M, Li Z, Mavros Y, Sachdev PS, Valenzuela MJ. Hippocampal plasticity underpins long-term cognitive gains from resistance exercise in MCI. Neuroimage Clin. 2020;25:102182. doi: 10.1016/j.nicl.2020.102182. Epub 2020 Jan 14. PMID 31978826
- [Background] Weterings S, Oppewal A, van Eeden FMM, Hilgenkamp TIM. A resistance exercise set for a total body workout for adults with intellectual disabilities, a pilot study. J Appl Res Intellect Disabil. 2019 May;32(3):730-736. doi: 10.1111/jar.12552. Epub 2018 Dec 10. PMID 30536559